CLINICAL TRIAL: NCT04410757
Title: Point of Care Ultrasound Evaluation in the Post-Anesthesia Unit- A Collaborative Observational Study Between UCLA and Loma Linda University Medical Centers
Brief Title: Point of Care Ultrasound Evaluation in the Post-Anesthesia Unit
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Davinder Ramsingh, MD, Director of Clinical Research, Loma Linda University
Other Study IDs: 5180035
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Hypotension; Hypoxemia; Altered Mental Status; Urine Output Low; Chest Pain
MeSH Terms: conditions — Hypotension; Hypoxia; Oliguria; Chest Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Point of Care Ultrasound (POCUS) group: When the provider in charge of covering the post-anesthesia care unit, they would apply POCUS examinations in their PACU assessment as per the study protocol of hypotensive and hypoxic events.
- No Point of Care Ultrasound (POCUS) group: When the provider in charge of covering the post-anesthesia care unit, they would apply routine bedside examination techniques in their PACU assessment as per the study protocol of hypotensive and hypoxic events.

SUMMARY:
The purpose of this observational research study is to examine how point-of care ultrasound affects the workup and management of perioperative complications for specific clinical scenarios of low blood pressure (hypotension), low blood oxygen (hypoxemia), in the post- anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Patients in the post-anesthesia care unit with the following events
* Mean arterial blood pressure <60 mmHg or <20% of pre-operative baseline mean arterial blood pressure,) hypoxemia (pulse oximetry saturation <95% or Pao2 <80), altered mental status, decreased urine output, chest pain/EKG changes, or to confirm endotracheal Lube placement.

Exclusion Criteria:

* Patients who are not able to have a point of care ultrasound examination in the post anesthesia recovery area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient or outpatient subjects from the age 18 and above with no maximum age limit admitted in the post-anesthesia care unit (PACU) that experienced a hypoxic or hypotensive event and were examined by a physician.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
post anesthesia care (PACU) unit length of stay (minutes) | during year of the study enrollment
  The primary outcome marker for the study was post anesthesia care (PACU) unit length of stay (minutes), with a hypothesis that patients receiving a POCUS examination for the cardiovascular or pulmonary event would have a shorter PACU LOS.

SECONDARY OUTCOMES:
number of diagnosis before and after assessment | during of the study enrollment
  Additional markers include a POCUS report completed by the performing attending anesthesiologist that included POCUS findings and the number of potential diagnoses to explain the acute event (hypoxia and/or hypotension) before and after the POCUS exam was performed..

CONTACTS AND LOCATIONS:
Overall Officials: Davinder Ramsingh, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Department of Anesthesiology, Loma Linda, California, United States

REFERENCES:
- [Background] Ramsingh D, Rinehart J, Kain Z, Strom S, Canales C, Alexander B, Capatina A, Ma M, Le KV, Cannesson M. Impact assessment of perioperative point-of-care ultrasound training on anesthesiology residents. Anesthesiology. 2015 Sep;123(3):670-82. doi: 10.1097/ALN.0000000000000776. PMID 26181338
- [Background] Canty DJ, Royse CF, Kilpatrick D, Bowman L, Royse AG. The impact of focused transthoracic echocardiography in the pre-operative clinic. Anaesthesia. 2012 Jun;67(6):618-25. doi: 10.1111/j.1365-2044.2012.07074.x. Epub 2012 Feb 21. PMID 22352785
- [Background] Ford JW, Heiberg J, Brennan AP, Royse CF, Canty DJ, El-Ansary D, Royse AG. A Pilot Assessment of 3 Point-of-Care Strategies for Diagnosis of Perioperative Lung Pathology. Anesth Analg. 2017 Mar;124(3):734-742. doi: 10.1213/ANE.0000000000001726. PMID 27828799
- [Background] Haskins SC, Desai NA, Fields KG, Nejim JA, Cheng S, Coleman SH, Nawabi DH, Kelly BT. Diagnosis of Intraabdominal Fluid Extravasation After Hip Arthroscopy With Point-of-Care Ultrasonography Can Identify Patients at an Increased Risk for Postoperative Pain. Anesth Analg. 2017 Mar;124(3):791-799. doi: 10.1213/ANE.0000000000001435. PMID 27551733
- [Background] Perlas A, Van de Putte P, Van Houwe P, Chan VW. I-AIM framework for point-of-care gastric ultrasound. Br J Anaesth. 2016 Jan;116(1):7-11. doi: 10.1093/bja/aev113. Epub 2015 May 7. No abstract available. PMID 25951832
- [Background] Shokoohi H, Boniface KS, Pourmand A, Liu YT, Davison DL, Hawkins KD, Buhumaid RE, Salimian M, Yadav K. Bedside Ultrasound Reduces Diagnostic Uncertainty and Guides Resuscitation in Patients With Undifferentiated Hypotension. Crit Care Med. 2015 Dec;43(12):2562-9. doi: 10.1097/CCM.0000000000001285. PMID 26575653